CLINICAL TRIAL: NCT04396171
Title: Association of Probable Bruxism With Periodontal Status: A Cross Sectional Study
Brief Title: Association of Probable Bruxism With Periodontal Status
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Mehtap Bilgin Çetin, Dr. Mehtap Bilgin Çetin, Baskent University
Other Study IDs: MBCetin
Record Dates: First submitted 2020-05-16; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Probable bruxism(+)
- Probable bruxism(-)

SUMMARY:
This cross-sectional study was conducted to assess i) the prevalence of probable bruxism ii) the association between probable bruxism and periodontal status.The age, gender, education level, tooth loss, presence of probable bruxism and periodontal status of patients were evaluated. Periodontal statuses of the participants were defined according to the American Association of Periodontology/European Federation of Periodontology, 2017 consensus and assessment of probable bruxism was performed according to the 2018 consensus report on the assessment of bruxism.

DETAILED DESCRIPTION:
This cross-sectional study was conducted to assess i) the prevalence of probable bruxism ii) the association between probable bruxism and periodontal status dental examination, all participants completed a standardized questionnaire. Sociodemographic findings comprised age, gender and educational level. Periodontal statuses of the participants were defined according to the American Association of Periodontology/European Federation of Periodontology, 2017 consensus. Participants were diagnosed with periodontitis if interdental clinical attachment loss (AL) was detected at ≥2 non-adjacent teeth, or buccal or oral AL was ≥3 mm with probing depth >3 mm was detected at ≥2 teeth. 12 In addition number of missing teeth is recorded.Assessment of probable bruxism was performed according to the 2018 consensus report on the assessment of bruxism.Presence of masticatory muscle hypertrophy, temporomandibular joint pain, indentations on the tongue or lip and/or a linea alba on the inner cheek, damage to the dental hard tissues (eg, cracked teeth), mechanical wear of the teeth (ie, attrition), repetive failures of restorative work/prosthodontics constructions were examined in clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years and older

Exclusion Criteria:

* age under 18 years,
* edentulous patients,
* not interested to participate in this study.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who applied to Department of Periodontology, Baskent University were included into the study.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
probable bruxism | 5 minutes
  Assessment of probable bruxism was performed according to the 2018 consensus report on the assessment of bruxism. For this purpose clinical inspection, one of the non-instrumental approaches, was used to evaluate the clinical features of bruxism. Presence of masticatory muscle hypertrophy, temporomandibular joint pain, indentations on the tongue or lip and/or a linea alba on the inner cheek, damage to the dental hard tissues (eg, cracked teeth), mechanical wear of the teeth (ie, attrition), repetive failures of restorative work/prosthodontics constructions were examined in clinical evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University,Department of Dentistry, Ankara, Turkey (Türkiye)